CLINICAL TRIAL: NCT01052649
Title: Gene Expression Monitoring of Peripheral Blood Mononuclear Cells Subpopulations (CD4+ Cells, CD56+ Cells and CD4+CD25+ Cells) and Immunological Status and Metabolome Defining of Healthy Population
Brief Title: Gene Expression Monitoring of Mononuclear Cells (MNC) Subpopulations and Immunological Status and Metabolome Defining of Healthy Population
Status: Completed | Type: Observational
Sponsor: Blood Transfusion Centre of Slovenia (Other Government)
Other Study IDs: MNC -1-4
Record Dates: First submitted 2009-07-24; First posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-07

CONDITIONS: Gene Expression; Metabolomics; Immunological Status
Keywords: MNC subpopulations; Gene Expression; Metabolomics; Immunological Status
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling

SUMMARY:
Study on healthy volunteers is focusing on analysis of transcriptome profile fluctuations in healthy population in three mononuclear cell types (CD4+ cells, CD56+ cells and CD4+CD25+ cells)and should provide a reference for comparison with transcriptomic data of any disease state.Furthermore, metabolome and immunological status are defined on same samples.

ELIGIBILITY:
Inclusion Criteria:

* age: 20-70 years
* healthy

Exclusion Criteria:

* acute or chronic diseases
* pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy population
Sampling Method: Probability Sample
Dates: Start 2008-08

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Transfusion Centre of Slovenia, Ljubljana, Ljubljana, Slovenia